CLINICAL TRIAL: NCT01264198
Title: The Role of Resistance Training in Non Alcoholic Fatty Liver Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Prof. Ran Oren, Tel-Aviv Sourasky Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TASMC-10-RO-330-CTIL
Record Dates: First submitted 2010-07-06; First posted 2010-12-21 (Estimated); Last update posted 2014-03-27 (Estimated); Status verified 2010-12

CONDITIONS: NAFLD (Non-Alcoholic Fatty Liver Disease); Resistance Training
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Stretching Exercises (Sham Comparator): The patients will perform twice weekly home based static stretching workout.
  Interventions: Behavioral: Resistance Training
- Resistance Training (Experimental): The patients will perform twice weekly supervised RT for 3 months
  Interventions: Behavioral: Resistance Training

INTERVENTIONS:
Behavioral: Resistance Training — Supervised Resistance Training

SUMMARY:
The aim of the study is to evaluate the effect of RT on clinical and metabolic parameters in patients with NAFLD.

DETAILED DESCRIPTION:
Background: Non Alcoholic Fatty Liver Disease (NAFLD) is the most prevalent liver disease in developed countries with a prevalence rate of 20-30 % of adults. About 10-25% of these individuals are estimated to meet the current diagnostic criteria for Non Alcoholic Steatohepatitis (NASH) and some may progress to Cirrhosis and liver failure. NAFLD is now recognized as the hepatic manifestation of the metabolic syndrome. Recent data shows that NAFLD might also predict the tendency to develop diabetes mellitus and coronary artery disease. The drug of choice for NAFLD is yet to be found. The recommended treatment of NAFLD includes weight reduction and Physical Activity (PA), but the data of the effect of Resistance Training (RT) PA on NAFLD is scant.

Aim of the study: To evaluate the effect of RT on clinical and metabolic parameters in patients with NAFLD. Study design: Randomized Clinical Trial. Patients will be randomly allocated to 2 arms (intervention and control). The intervention arm will perform RT, whereas control arm will be advised to perform home stretching. Medical examination will be performed at week 0 (baseline) and at week 13 using uniform protocols.

ELIGIBILITY:
Inclusion Criteria:

* Ultrasound diagnosed fatty liver.

Exclusion Criteria:

* Presence of HBsAg or anti-HCV antibodies (will be obtained from blood tests at the liver clinic).
* Patients with known diabetes treated with antidiabetic medications.
* Patients with known kidney disease, CHD, lung disease, inflammatory bowel disease.
* Excessive alcohol consumption ≥ 30 g/day in men or 20 g/ day in women.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 82 (Actual)
Dates: Start 2010-12; Primary Completion 2012-09 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
The HRI value will be reduced in the intervention arm as compared to the The The change in Hepato-Renal Index (HRI) evaluated by ultrasound (US). | week 0 and week 13

CONTACTS AND LOCATIONS:
Overall Officials: Ran Oren, MD, Principal Investigator — Tel-Aviv Sourasky Medical Center
Locations (1):
- Tel Aviv Sourasky Medical center, Tel Aviv, Israel

REFERENCES:
- [Derived] Zelber-Sagi S, Azar S, Nemirovski A, Webb M, Halpern Z, Shibolet O, Tam J. Serum levels of endocannabinoids are independently associated with nonalcoholic fatty liver disease. Obesity (Silver Spring). 2017 Jan;25(1):94-101. doi: 10.1002/oby.21687. Epub 2016 Nov 15. PMID 27863097